CLINICAL TRIAL: NCT04307095
Title: Incidence of Postoperative Hypothermia and Associated Factors in Adult Patients Undergoing Surgery in Siriraj Hospital
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Associate Professor, Siriraj Hospital
Other Study IDs: IRB889
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hypothermia Following Anesthesia
Keywords: Postoperative hypothermia; Patient warming; Inadvertent hypothermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inadvertent postanesthetic hypothermia is unintentional drop in core body temperature <36C (96.8F) immediately following an operation, caused by multiple factors, and had lead to negative outcomes. In our institute, a study in 2011 reported an incidence of postoperative hypothermia in PACU of 45.4% (95% CI 39.61%- 51.23%). After that, various interventions aimed to prevent perioperative hypothermia were implemented. This study is initiated to determine the incidence of postoperative hypothermia and associated factors of postoperative hypothermia in adult patients underwent surgery at Siriraj hospital.

DETAILED DESCRIPTION:
Inadvertent postanesthetic hypothermia is unintentional drop in core body temperature <36C (96.8F) immediately following an operation, which is a common problem in post anesthesia care unit (PACU). It has been implicated in negative outcomes in surgical patients, including prolonged effects of intraoperative anesthetic medication, increased insulin resistance, postoperative morbidity, delayed surgical wound healing; and prolonged stay in the recovery room and hospital1-7.

In the operating room (OR), patients have to expose to a low ambient temperature with little or no clothing, evaporation from the surgical area, an irrigated fluid in surgical area; and an administration of intravenous fluids. Moreover, many anesthetic agents have an influence on the autonomic thermoregulatory mechanism which causes vasodilatation. All these factors promote patients' unintentional loss of heat and cause hypothermia.

Even of a lot of efforts to keep patients warm intraoperatively and minimize hypothermia including optimizing ambient OR temperature and using of various warming devices, the incidences of postoperative hypothermia in PACU are still high with the reported magnitude ranges from 50%- 90%7. In Siriraj hospital, a study in 2011 reported an incidence of postoperative hypothermia in PACU of 45.4% (95% CI 39.61%- 51.23%)8. After that, various interventions aimed to prevent perioperative hypothermia were implemented such as maintaining the ambient room temperature of an OR; warming intravenous fluids, blood products, and irrigants; heated, humidified anesthetic gases; and using warming blankets, forced-air warming, layering drapes and head wraps. This study is initiated to determine the incidence of postoperative hypothermia and associated factors of postoperative hypothermia in adult patients underwent surgery at Siriraj hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years undergoing surgery with anesthesia service
* Stay at Postanesthetic care unit of Syamindra building, fifth floor, Siriraj hospital

Exclusion Criteria:

* Procedure performed under local anesthesia
* Patients with missing data of temperature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of age more than 18 years old who undergoing anesthesia and surgery in Siriraj hospital.
Sampling Method: Non-Probability Sample
Enrollment: 742 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Body temperature | 1 min
  Body temperature after admit in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Faculty of medicine Siriraj hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mauermann WJ, Nemergut EC. The anesthesiologist's role in the prevention of surgical site infections. Anesthesiology. 2006 Aug;105(2):413-21; quiz 439-40. doi: 10.1097/00000542-200608000-00025. No abstract available. PMID 16871076
- [Background] Panagiotis K, Maria P, Argiri P, Panagiotis S. Is postanesthesia care unit length of stay increased in hypothermic patients? AORN J. 2005 Feb;81(2):379-82, 385-92. doi: 10.1016/s0001-2092(06)60420-1. PMID 15768547
- [Background] Wartzek T, Muhlsteff J, Imhoff M. Temperature measurement. Biomed Tech (Berl). 2011 Oct;56(5):241-57. doi: 10.1515/BMT.2011.108. PMID 21988157
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Background] Insler SR, Sessler DI. Perioperative thermoregulation and temperature monitoring. Anesthesiol Clin. 2006 Dec;24(4):823-37. doi: 10.1016/j.atc.2006.09.001. PMID 17342966
- [Background] Kiekkas P, Poulopoulou M, Papahatzi A, Souleles P. Effects of hypothermia and shivering on standard PACU monitoring of patients. AANA J. 2005 Feb;73(1):47-53. PMID 15727284
- [Derived] Wongyingsinn M, Pookprayoon V. Incidence and associated factors of perioperative hypothermia in adult patients at a university-based, tertiary care hospital in Thailand. BMC Anesthesiol. 2023 Apr 25;23(1):137. doi: 10.1186/s12871-023-02084-2. PMID 37098492